CLINICAL TRIAL: NCT06530238
Title: Comparative Study Between Russian And Exercise in Subjects With Flexible Flatfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physical Therapy 3
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Flat Feet
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Experimental): Russian current
  Interventions: Procedure: Russian Currents
- Group (B) (Active Comparator): Exercise
  Interventions: Procedure: Russian Currents

INTERVENTIONS:
Procedure: Russian Currents — Currents are delivered in rectangular bursts. The electrode placement will be at the Tibialis Posterior muscle. Treatment will be given for 10 minutes, 30 minutes during the 3 consecutive days / 4 weeks.

SUMMARY:
The prevalence of flexible flat foot was 13.6% in adults a cross-sectional Study (for males-12.8%; for females-14.4%).18-21-year-old Indian adults. This trial aims to compare between the effects of Russian current for tibialis posterior muscle and comprehensive exercise alone in subjects suffering from flexible flat foot on quality of life, ROM, strength of tibialis posterior and foot posture

ELIGIBILITY:
Inclusion Criteria:

* The patient's age ranges from 20 to 25 years.
* Both genders.
* patients suffering from symptomatic flat foot

Exclusion Criteria:

* Rigid flatfoot.
* Pregnancy and lactation.
* recent fracture and fixation.
* genu valgus.
* cardiac pacemaker.
* inflammatory disorders / rheumatoid arthritis.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
ROM (inversion and eversion). | 4 weeks
  Universal goniometer to assess the ROM (inversion and eversion) of the subtalar joint for each patient
Foot Posture Index (FP1-6) | 4 weeks
  The FPI-6 is a novel method of rating foot posture using set criteria and a simple scale and is a quick, reliable diagnostic tool.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Nouran adam, Minya, Select Region
  - Deraya university, Minya